CLINICAL TRIAL: NCT01418833
Title: Preliminary Experience of Routine Voriconazole Therapeutic Drug Monitoring (TDM) in a Tertiary Care Centre.
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Ap.r Kim Vanstraelen, Hospital Pharmacist, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: ML7258
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Patients Treated With Voriconazole
Keywords: voriconazole; therapeutic drug monitoring; plasma levels; dose adjustment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The first goal of this study is to map all the subtherapeutic, therapeutic and supratherapeutic voriconazole plasma levels in the University Hospitals Leuven. The second objective is to optimize and validate guidelines for dose modifications in patients with too low or high plasma concentrations and to investigate if the same guidelines can be used in different patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with voriconazole
* at least 1 voriconazole plasma level measured during therapy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with voriconazole, in whom at least 1 voriconazole plasma level was determined
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Voriconazole plasma levels during routine intravenous and oral therapy | trough levels every 4 days after start or dose adjustment of voriconazole

CONTACTS AND LOCATIONS:
Overall Officials: Kim Vanstraelen, R.Ph., Principal Investigator — Catholic University of Leuven, Faculty of Pharmacy, division Hospital Pharmacy
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium